CLINICAL TRIAL: NCT02882178
Title: Formal Consensus Method to Evaluate the Conformity of Prescription of a Recently Approved Chemotherapy Treatment in an Observatory Study
Brief Title: Consensus Method to Evaluate the Conformity of Prescription of a Chemotherapy
Acronym: CABOBS
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Sanofi (Industry); GECEM (Industry)
Responsible Party: Sponsor
Other Study IDs: IB2012-CABOBS
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; cabazitaxel; consensus; conformity; prescription; conditions of use
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Cabazitaxel is a second line chemotherapy drug recently approved for the treatment of metastatic castration-resistant prostate cancer. To investigate whether the precautions for the use of cabazitaxel (contraindications, hepatic function, premedication for hypersensitivity, prophylactic treatments, dose and dose adjustment, as well as conditions of administration) are respected in routine practice, an observational cohort study will be implemented in 32 oncology centres of South-West region of France (CABOBS study). The primary objective of this cohort is to evaluate the conformity of cabazitaxel prescriptions with the Summary of Product haracteristics (SPC) in clinical practice (indications and monitoring methods) and according to the conditions of use. Panel of experts were convened to assess the conformity of prescription of cabazitaxel with a Delphi consensus method. The Delphi method is most suited to areas where a limited number of evidences are available to enable a recommendation or guidelines to be drawn. Moreover, all the evaluated items came from an official document provided by the EMA, the SPC of cabazitaxel. Thus, it is expected from the experts to select the most relevant items. In the frame of the CABOBS study, this method will allow to select items of the SPC list according to their importance, and to define the primary objective of conformity to cabazitaxel conditions of use.

DETAILED DESCRIPTION:
For metastatic castration-resistant prostate cancer (mCRPC) patients, treatment usually consists in a first line chemotherapy with docetaxel followed by a second line treatment with either second generation hormonal therapies (abiraterone acetate or enzalutamide) or the new taxane derivative cabazitaxel. Cabazitaxel (Jevtana) is a semi-synthetic taxane with a mechanism of action different to that of docetaxel and paclitaxel. It is an antineoplastic agent that stabilises the microtubules network via its binding to tubulins and the inhibition of microtubules disassembly. Cabazitaxel has demonstrated a broad spectrum of antitumour activity against advanced human tumours xenografted in mice. It is active in docetaxel-sensitive tumours and in tumour models resistant to chemotherapy, including docetaxel. The efficacy of cabazitaxel has been demonstrated in the pivotal clinical trial TROPIC, a randomized, open-label, phase III study that compared cabazitaxel (n = 378) to mitoxantrone (n = 377), both associated with prednisone or prednisolone in patients with hormone-refractory metastatic prostate cancer previously treated with a docetaxel containing regimen. The median overall survival (OS) was significantly increased in the cabazitaxel-treated group compared to the mitoxantrone-treated group. Most common adverse event that can lead to a treatment discontinuation are haematological (neutropenia 82%), gastrointestinal (diarrhoea 6%) and general disorders (asthenia 5%). A recent study analysed the data of the TROPIC study on efficacy and toxicity observed in the subgroup of patients included in French centres. These results are comparable to those reported for the overall population and the safety profile remains favourable without any toxic death related to cabazitaxel.

Following TROPIC trial, cabazitaxel (in combination with prednisone or prednisolone) was approved by the U.S. Food and Drug Administration (FDA) on June 2010 and by the European Medicines Agency (EMA) on March 2011 for the treatment of hormone-refractory prostate cancer. In France cabazitaxel was approved in 2012 but made available only in 2014.

To investigate whether the precautions for the use of cabazitaxel (contraindications, hepatic function, premedication for hypersensitivity, prophylactic treatments, dose and dose adjustment, as well as conditions of administration) are respected in routine practice, an observational cohort study will be implemented in 32 oncology centres of South-West region of France (CABOBS study). The primary objective of this cohort is to evaluate the conformity of cabazitaxel prescriptions with the Summary of Product Characteristics (SPC) in clinical practice (indications and monitoring methods) and according to the conditions of use.

Based on the SPC, Specifications for prescription include 26 items divided into "baseline" (14) criteria and "cycle 2" (12) criteria, which include requirements for the second and all following cycles. Because of such high number of specific items, strict adherence to prescription indications might be unsatisfactory or not appropriate from the clinical point of view, each criterion has a different relevance on the appropriateness of prescription; therefore, it is necessary to select the criteria based on their relevance and according to the opinion of the clinical experts.

For this purpose, two independent panels of experts in the field of uro-oncology, one French panel and a European panel from EORTC, were solicited in order to define the importance of each criterion of the SPC and to allow a qualitative assessment of conformity using a formal consensus method.

Consensus methods provide means of synthesising information and compare contradictory opinions or evidences on a specific issue. Their purpose is to assess the extent of agreement and to resolve disagreement among a group of selected individuals by identifying and selecting, through iterative ratings with feedback, specific points on which there is disagreement or uncertainty.

The Delphi method, a consensus method which originated in 1948, is an attempt to obtain expert opinion in a systematic manner. The survey is conducted over "rounds" in which questionnaires are administered to the experts individually and anonymously. After each round, the results are listed and reported to the group. A Delphi is considered complete when there is a convergence of opinion. In a modified Delphi usually a predefined number of rounds and a final round, in which experts meet to resolve and summarise the results of the consensus, are held.

The Sponsor relied on the Delphi method as it is most suited to areas where a limited number of evidences are available to enable a recommendation or guidelines to be drawn. Moreover, all the evaluated items came from an official document provided by the EMA, the SPC of cabazitaxel. Thus, it is expected from the experts to select the most relevant items. In the frame of the CABOBS study, this method will allow to select each of the 26 items of the SPC list according to their importance, and to define the primary objective of conformity to cabazitaxel conditions of use.

ELIGIBILITY:
Eligibility criteria for the experts involved in the consensus process:

1. experts in uro-oncology solicited within the French GETUG's group (Groupe d'Etude des Tumeurs Uro-Génitales)
2. experts in uro-oncology solicited within the EORTC GU group for the second panel of experts.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Experts of the consensus process
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HOUEDE Nadine, Principal Investigator — Institut Bergonié

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Houede N, Leutenegger E, Lomma M, Bellera C. Formal consensus method to evaluate the conformity of prescription of a recently approved chemotherapy treatment in an observatory study. PLoS One. 2015 Apr 2;10(4):e0123035. doi: 10.1371/journal.pone.0123035. eCollection 2015. PMID 25837603

RESULTS

PARTICIPANT FLOW:
Groups:
- Experts of the Consensus Process: Experts involved in the consensus process
Period: Overall Study
Arm/Group | Experts of the Consensus Process
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experts of the Consensus Process
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  > 18 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 18

OUTCOME MEASURES:

1. Primary Outcome: Items to Define Conformity to Cabazitaxel Conditions of Use
Description: Items selected by the consensus process to assess the conformity of prescription of cabazitaxel based on the the 26 items included in the Summary of Product Characteristics (SPC). Two independent panels of experts in the field of uro-oncology, one French panel and a European panel from the Genito-Urinary group of the European Organization for Research and Treatment of Cancer (EORTC-GU), were solicited in order to define the importance of each criterion of the SPC and to allow a qualitative assessment of conformity using a formal consensus method. The purpose of consensus methods is to assess the extent of agreement and to resolve disagreement among a group of selected individuals by identifying and selecting, through iterative ratings with feedback, specific points on which there is disagreement or uncertainty. We relied on the Delphi method as it is most suited to areas where a limited number of evidences are available to enable a recommendation or guidelines to be drawn.
Time Frame: Baseline
Measure: Number; unit: items
Arm/Group | Experts of the Consensus Process
Number analyzed (Participants) | 18
items | 11

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Experts of the Consensus Process
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes